CLINICAL TRIAL: NCT06640218
Title: The Effect of Eddy Sonic Versus AF Max Activation of Bio-ceramic Sealer on Post-operative Pain in Teeth with Symptomatic Irreversible Pulpitis with Apical Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Youssef Abd El Hameed Mohamed Ahmed, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUE-REC code (17)/7/2024
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Irreversible Pulpitis with Apical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bio-ceramic sealer activation with Eddy sonic before obturation (Active Comparator): cleaning and shaping the root canals and Well Root bio ceramic sealer activation using Eddy sonic before obturation
  Interventions: Device: sealer activation with Eddy sonic and AF max
- bio-ceramic sealer activation with AF max before obturation (Active Comparator): cleaning and shaping the root canals and Well Root bio ceramic sealer activation using AF max before obturation
  Interventions: Device: sealer activation with Eddy sonic and AF max
- bio-ceramic sealer obturation without any activation (negative control) (Active Comparator): obturation of root canals with bio ceramic sealer directly without any activation
  Interventions: Other: without AF max or Eddy sonic sealer activation

INTERVENTIONS:
Device: sealer activation with Eddy sonic and AF max — activation of sealer after cleaning and shaping, before the obturation
  Arms: bio-ceramic sealer activation with AF max before obturation; bio-ceramic sealer activation with Eddy sonic before obturation
Other: without AF max or Eddy sonic sealer activation — sealer without activation
  Arms: bio-ceramic sealer obturation without any activation (negative control)

SUMMARY:
The aim of endodontic therapy for an inflamed tooth is to eliminate the source of inflammation. Relieving pain depends on the effectiveness of root canal therapy.3

Postoperative pain in endodontic treatments, affecting 3-58% of patients, is often caused by peri-radicular tissue injuries. Understanding these factors helps professionals select methods and supplies to minimize discomfort.

30 patients will be divided into 3 groups according to the method of activation (10 par ticipants/each). participants will be recruited from the postgrad clinic of the endodontic department faculty of oral and dental medicine, Future University in Egypt Patients with mature mandibular first permanent molar with irreversible pulpitis with apical periodontitis Intervention 1: bio-ceramic sealer activation with Eddy sonic Intervention 2: bio-ceramic sealer activation with AF max Control/Comparator: bio-ceramic sealer without activation The study aims to evaluate the effect of Eddy Sonic and AF max activation of bio-ceramic sealer on postoperative pain in mandibular first molars with symptomatic irreversible pulpitis with apical periodontitis

ELIGIBILITY:
Inclusion Criteria:

* Age range is from 18 to 40 years old.
* No sex predilection
* Patients seeking root canal treatment.
* restorable teeth.
* Positive patient acceptance for participating in the study.
* patients able to sign informed consent.
* Systematically healthy patient (ASA I, Il).
* Patient who can understand the numerical rate scale and sign an informed consent.
* Mandibular first molar teeth with pain on bite or percussion
* Preoperative sharp (moderate or severe) pain.
* Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).
* widening in periodontal membrane space in radiographic appearance.

Exclusion Criteria:

* Patients with American Association of Anesthesiologists (ASA) classifications other than ASA 1 & Il
* Patients who have already ingested preoperative medication, such as analgesics, non-steroidal, or steroidal anti-inflammatory drugs, within 12 hours of the start of treatment.
* This was done to prevent any misinterpretation of the diagnosis or post-treatment pain severity, as these drugs substantially lower post-endodontic pain (Jorge-Arajo et al.,2018).
* Patients with NSAID allergy.
* Patients having two or more adjacent teeth needing root canal therapy
* Pregnant patients.
* Patients with bleeding disorder.
* Patients with long-term corticosteroid use.
* Teeth having:

  * Necrotic pulp.
  * History or presence of swelling or fistulous tract.
  * Acute/chronic periapical abscess.
  * Mobility more than grade 1.
  * Pocket depth of more than 5mm
  * No possible restorability.
  * Previous root canal treatment.
  * Periapical radiolucency.
  * External or internal resorption
  * Vertical root fracture.
* TMJ problems, bruxism, clenching or traumatic occlusion.
* Inability to understand and perform the given instructions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
post-operative pain after root canal treatment with sealer activation by AF max and Eddy sonic activation in comparison to without sealer activation | Immediately after obturation 6-12-24 and 48 hours post-operative
  measuring post-operative pain by Numerical rate scale and pain level will be assigned to one of 4 categorical scores: None (0); Mild (1-3); Moderate (4-6); Severe (7-10).

SECONDARY OUTCOMES:
Number of analgesic tablets taken after endodontic treatment | Up to 48 hours post-operative pain
  measuring number of analgesic tablets taken after endodontic treatment by counting

OTHER OUTCOMES:
radiographic presence or absence of sealer extrusion | Immediately after obturation
  detecting lateral and periapical sealer extrusion through postoperative periapical radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided